CLINICAL TRIAL: NCT02566811
Title: A Randomised Trial of Non-selective Versus Selective Adjuvant Therapy in High Risk Apparent Stage 1 Endometrial Cancer
Brief Title: Selective Targeting of Adjuvant Therapy for Endometrial Cancer (STATEC)
Acronym: STATEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of funding by CR UK due to poor recruitment
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0630
Record Dates: First submitted 2015-09-22; First posted 2015-10-02 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-06

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal surgery with lymphadenectomy (Experimental): Patients will receive a hysterectomy and bilateral salpingo-oophorectomy (BSO)* with lymph node dissection to determine whether lymph nodes are positive or negative:
  Positive: patients will receive systemic adjuvant treatment to include chemotherapy Negative: patients will receive vaginal brachytherapy only
  Patients will then be followed up, to include assessment of adverse events and quality of life.
  *There is an option for patients to be randomised following a pre-trial hysterectomy and BSO. If randomised to this arm, the lymph node dissection will be performed as a separate procedure.
  Interventions: Procedure: Abdominal surgery; Procedure: Lymphadenectomy
- Abdominal surgery, no lymphadenectomy (Active Comparator): Patients will receive a hysterectomy and bilateral salpingo-oophorectomy (BSO)*. Patients will receive systemic adjuvant treatment to include chemotherapy.
  Patients will then be followed up, to include assessment of adverse events and quality of life.
  *There is an option for patients to be randomised following a pre-trial hysterectomy and BSO. If randomised to this arm, no further surgery will be given and the patient will proceed to receive systemic adjuvant treatment to include chemotherapy.
  Interventions: Procedure: Abdominal surgery

INTERVENTIONS:
Procedure: Abdominal surgery — Hysterectomy defined as an extrafascial hysterectomy whereby the cervix is removed completely but no radical dissection of the parametria is required
Procedure: Lymphadenectomy — Bilateral pelvic and para-aortic lymph node dissection
  Arms: Abdominal surgery with lymphadenectomy

SUMMARY:
The primary aim of this trial is to determine whether lymphadenectomy, used to restrict adjuvant therapy (other than vaginal brachytherapy) to node positive women, results in a non-inferior survival as compared to adjuvant therapy given to all women with high risk apparent stage 1 endometrial cancer.

DETAILED DESCRIPTION:
Results from this trial have the potential to change practice whatever the results: either lymphadenectomy will become recommended practice if a non-inferior outcome is obtained; otherwise the procedure can be safely abandoned.

Secondary Objectives

* Disease-free, endometrial cancer-event free and endometrial cancer-specific survival
* Distribution of pelvic and extra-pelvic relapse
* Cost effectiveness
* Surgical adverse events

There are also two sub-studies:

1. Quality of life - all patients i. Describe the trajectory of key patient reported outcomes (PROs) from baseline up to 5 years post-surgery ii. Compare the specific PRO domains between the trial arms at several specific time points iii. Determine the proportion of women in each trial arm reporting long-term symptoms after treatment as measured by the symptom-specific subscales of the measures (gastrointestinal symptoms, urological symptoms, attitude to disease and treatment, vaginal symptoms, lymphoedema) iv. Determine the correlation between physician rating (CTCAE v4.03) and patient-report (corresponding PRO subscale) for various symptoms reported by both physicians and patients v. Assess the correlation between self-assessed lymphoedema (Self-report lower-extremity lymphoedema screening questionnaire) and the lymphoedema subscale of the Quality of Life Questionnaire-Endometrial Cancer Module (QLQ-EN24)

   We hypothesise that quality of life will be better in patients in the lymphadenectomy arm because a considerable proportion will be spared systemic adjuvant treatment, from which they may not benefit.
2. Sentinel lymph node (SLN) - optional for Arm 1 patients

The aim of this sub-study is to assess SLN status in comparison with the overall lymph node status after full lymph node dissection (LND), and so determine whether SLN is as accurate as systematic node dissection.

i. We aim to determine the diagnostic performance of the SLN procedure compared to the gold standard of LND ii. To evaluate whether SLN status is a prognostic marker of survival iii. To model patient relapse and survival based on low volume micro-metastatic (LVM) and individual tumour cell (ITC) status

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high risk apparent International Federation of Gynecology and Obstetrics (FIGO) stage I endometrial cancer according to one of the following criteria. Confirmation must be based on either diagnostic endometrial sampling or hysterectomy and BSO specimen if randomisation occurring after hysterectomy and BSO:

  1. FIGO grade 3 endometrioid or mucinous carcinoma
  2. High grade serous, clear cell, undifferentiated or dedifferentiated carcinoma or mixed cell adenocarcinoma or carcinosarcoma
* Surgery to be performed ≤ 5 weeks after randomisation in patients randomised prior to hysterectomy and BSO. Patients randomised after hysterectomy and BSO must have undergone hysterectomy and BSO ≤ 28 days prior to randomisation. Patients randomised after hysterectomy and BSO who are allocated lymphadenectomy must undergo lymphadenectomy ≤ 5 weeks after randomisation
* Written informed consent
* No prior anticancer therapy for endometrial cancer
* Eastern Cooperative Oncology Group (EGOC) performance status 0-2
* Life expectancy > 3 months
* Age ≥ 16 years
* Adequate organ and bone marrow function
* Ability to undergo post-operative chemotherapy with or without radiotherapy
* Adjuvant treatment to commence ≤ 8 weeks after surgery
* Willingness and ability to complete Quality of Life questionnaires

Exclusion Criteria:

* Grossly enlarged node(s) of ≥ 10 mm short axis on baseline radiological imaging
* Invasion of the cervical stroma on baseline radiological imaging or obvious cervical disease on clinical examination
* Involvement of uterine serosa or metastatic disease seen outside the uterus on baseline radiological imaging
* Small cell carcinoma with neuroendocrine differentiation
* Concurrent anti-cancer therapy
* Previous malignancy < 5 years prior to randomisation or concurrent malignant disease with the exception of:

  1. carcinoma in situ of cervix
  2. non-melanoma skin cancer
  3. basal cell carcinoma
  4. melanoma in situ
* Women who are pregnant or lactating

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival
Endometrial cancer-event free survival | 5 years
  Endometrial cancer-event free survival
Endometrial cancer-specific survival | 5 years
  Endometrial cancer-specific survival
Pelvic and extra-pelvic relapse-free survival | 5 years
Cost effectiveness | 5 years
  Cost effectiveness
Surgical adverse events | 5 years
  Surgical adverse events

OTHER OUTCOMES:
Quality of life- Patient Reported Outcomes | 5 years
  Quality of life
Accuracy, sensitivity and specificity (i.e. diagnostic performance) of sentinel lymph node (SLN) assessment, and the ratio of sensitivity to false positive rate (called likelihood ratio) | 5 years
  Accuracy, sensitivity and specificity (i.e. diagnostic performance) of sentinel lymph node

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mould, Principal Investigator — University College London Hospital
Locations (1):
- University College Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No